Mindful Self-Compassion Training to Improve Retention, Job Satisfaction, and Attitudes toward Dementia among Long-Term Care Nursing Assistants:

Certified Nursing Assistants' Wellbeing

Analysis Overview. Analyses of the intervention's effectiveness will primarily comprise tests of changes to the outcome measures (see below) from baseline at three post-baseline timepoints: (a) post-intervention, (b) a 3-month follow-up, and (c) a 6-month follow-up. All outcomes were recorded at the same time points within the same self-report survey. Thus, overall, with baseline there were four data collection time points in the study. Secondarily, analyses will consider differences in effectiveness by comparing two intervention's two approaches: (a) the 20-hour intervention delivered in one NH and (b) the 6-hour intervention delivered in two additional NHs. In addition to outcome analyses, participants' univariate demographic and professional characteristics were calculated to describe the sample (not detailed). Missing data were not imputed, resulting in analyses using listwise deletion of participant observations without data at each time point and for each outcome. Statistical significance was set at p < 0.05 throughout (two-sided) and all analyses were conducted in Stata 16.1.

<u>Primary Outcome</u>. The primary outcome in the study was *Change in Intent to Leave Job*. The specific question asked of participants was "How likely is it that you will leave this job in the next year?" with intent to leave specifically being defined as a "Somewhat likely" or "Very likely" response (1 = Yes) versus a "Not at all likely" response (0 = No). The analysis of the primary outcome proceeded in two steps. First, the descriptive frequencies and percentages of "Yes" and "No" response were calculated for all participants at all four data collection time points to summarize the primary outcome across participants and time. Second, tests for the statistical significance of change from baseline was determined using three sets of McNemar's exact  $X^2$  tests compared baseline versus the three post-baseline time points. These tests were chosen as appropriate for the (a) non-parametric nature of the data and (b) paired nature of the comparison.

Secondary Outcomes. There were nine secondary outcome domains in the study: (a) mean Job Satisfaction Scale (JSS) score; (b) mean Approach to Dementia Questionnaire (ADQ) score; (c) mean Perceived Stress Scale (PSS) score; (d) mean PROMIS Depression Scale—Short Form (PROMIS) score, (e) mean subscale Maslach Burnout Inventory—Human Services Scale (MBI) scores; (f) mean total and subscale Self-Compassion Scale—Youth (SCS) scores; (g) Weekly Attendance; (h) Number of Days Per Week Spent in Out-of-Class Exercises; and (i) mean Satisfaction with Course score. Briefly, the JSS measured how satisfied participants were with at their job and included 3 individual items (Range: 0-18); the ADQ measured participants' attitudes toward NH residents with dementia and included 11 items (Range: 0-44); the PSS measured participants' stress and included 10 items (Range: 0-40); the PROMIS measured participants' depression levels and included 8 items (8-40); the MBI measured participants' burnout and included 20 items; the SCS measured participants' self-compassion and included 17 items; and the study-created Satisfaction with Course measure evaluated course-specific satisfaction and included 8 items. Rather than having a total score measuring burnout, the MBI featured 3 subscales related to Depersonalization, Emotional Exhaustion, and Reduced Personal Accomplishment constructs all with a range of 0.0-6.0. The SCS, meanwhile, featured a total score measuring self-compassion along with six subscales related to Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification constructs all with a total range of 1.0-5.0. All scales and sub-scales were summed into unweighted composites of individual items. Satisfaction with Course items all had five response options ranging from "Strongly disagree" (1) to "Strongly agree" (5). Weekly Attendance was defined as "% of intervention classes fully attended" with a possible score from > 0.0% to 100.0%. Meanwhile, Number of Days Per Week Spent in Out-of-Class Exercises was defined as "mean # of days per week over the course of the intervention spent out-of-class doing course mindfulness exercises" with a range from 1.0 to 7.0. The analysis of the secondary outcomes proceeded in three steps. First, the descriptive frequencies, percentages, means, and standard deviations of all measures were calculated for all participants at all four data collection time points to summarize the

secondary outcomes across participants and time. Second, tests for the statistical significance of change from baseline was determined using three sets of either (a) Wilcoxon sign-rank tests for continuous measures or (b) McNemar's exact  $X^2$  tests for nominal measures. These tests were chosen as appropriate for the (a) non-parametric nature of the data and (b) paired nature of the comparisons. Third, change from baseline stratified by intervention approach was determined by comparing the (a) change and (b) significance of the two sub-samples (i.e., 20-hour intervention, 6-hour intervention) for the (a) PSS, (b) PROMIS, and (c) total SCS scores.